CLINICAL TRIAL: NCT04382027
Title: Comparison of Pharmacokinetics of Omega-3 Fatty Acid Supplements in Monoacylglycerol or Ethyl Ester in Humans: a Randomized Controlled Trial.
Brief Title: Pharmacokinetics of Omega-3 Monoglycerides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Mélanie Plourde, Associate professor, Department of medicine, Geriatric service, Université de Sherbrooke
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PK1
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Healthy
Keywords: Omega-3 fatty acids; Vitamin K2; Bioavailability; Monoacylglycerol; Pharmacokinetic
MeSH Terms: interventions — Docosahexaenoic Acids; Vitamin K 2

STUDY DESIGN:
Intervention Model Description: Double-blind controlled-randomized pharmacokinetic (PK) pilot study with crossover design (10 men and 10 women), with a minimum of 6 days between treatments
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Neither the participant nor the research nurse will know the administration order of the different treatments administered. All plasma samples collected during the research project will be anonymized i.e. it will not be possible to identify the participant by his name since a number will be assigned to him. The code key linking the participant's name to his number will be stored, with access restricted to those designated by the principal investigator. The data file is also protected by a password.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Monoacylglycerol (Experimental): The participant will arrive fasted at Diex Recherche Sherbrooke. After installing a catheter and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive the omega-3 fatty acids as a unique dose of 3 g EPA + DHA in monoacylglycerol form + 45 mg vitamin K2. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma.
  Interventions: Dietary Supplement: Omega-3 + vitamin K2 (monoacylglycerol form)
- Ethyl ester (Active Comparator): The participant will arrive fasted at Diex Recherche Sherbrooke. After installing a catheter and drawing 5 mL of blood, the participants will be given one of the active comparator or the treatment. The choice of the treatment/comparator will be random. In this arm, the participant will receive the omega-3 fatty acids as a unique dose of 3 g EPA + DHA in ethyl ester form + 45 mg vitamin K2. The participant will consume this unique dose with a standardized breakfast. There will thereafter be blood sample collection over 24 h to evaluate the level of omega-3 fatty acids in the plasma.
  Interventions: Dietary Supplement: Omega-3 + vitamin K2 (ethyl ester)

INTERVENTIONS:
Dietary Supplement: Omega-3 + vitamin K2 (monoacylglycerol form) — The intervention is a randomized double bond cross over design testing the pharmacokinetics of a monoglyceride formulation compared to an ethyl ester form.
  Treatments are randomly assigned on days 0 and 7 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours. Each participant will perform the two treatments, with a minimum of 6 days between treatments.
  Arms: Monoacylglycerol
Dietary Supplement: Omega-3 + vitamin K2 (ethyl ester) — The intervention is a randomized double bond cross over design testing the pharmacokinetics of a monoglyceride formulation compared to an ethyl ester form.
  Treatments are randomly assigned on days 0 and 7 of the clinical study. Blood samples will be collected at time 0, 1, 2, 4, 5, 6, 8, 9, 10, 12 and 24 hours. Each participant will perform the two treatments, with a minimum of 6 days between treatments.
  Arms: Ethyl ester

SUMMARY:
North American diets have insufficient omega-3 fatty acid (n-3 FA) content. Consequently, they display low plasma concentrations of docosahexaenoic acid (DHA) and eicosapentaenoic acid (EPA), the two main long chain n-3 FA. A quick and easy way to increase the level of dietary n-3 FA is to take supplements. However, people report side effects in using the currently available supplements, such as gastrointestinal discomfort, nausea and gastric reflux; especially those where EPA and DHA are esterified as ethyl esters (EE). Moreover, EE supplements are less absorbed compared to other esterification forms, such as mono-, di- or triglycerides. The objective of this study was to test the pharmacokinetics of a new n-3 FA supplementation formulation rich in FAs esterified as monoacylglyceride (MAG).

DETAILED DESCRIPTION:
The growing presence on the North American as well as European market of food products enriched with fish oil as a source of polyunsaturated fatty acids (PUFA) omega-3 in the diet requires evaluation and comment. Research exploring health influence of the consumption of fish oil started in 1990 years. It was established that long-chain omega-3 PUFA (EPA C20:5 and DHA C22:6) has beneficial effect on human health. Fish oil is the main dietary source of long-chain omega-3 PUFA. Dietary recommendations suggest that the consumption of omega-3 PUFA should increase. The European Academy of Nutritional Sciences (EANS) and the United Kingdom dietary guidelines recommend a daily average intake of 0.2g of EPA plus DHA. In 2000, the Food and Drug Administration stated that the daily intake of EPA and DHA should increase up to 3.0 g per person in the form of fish oil, from food and dietary supplements. According to the World Health Organization recommendations for preventing cardiovascular diseases, one portion of fish should provide an equivalent of 200-500 mg of EPA and DHA. Due to the low fish consumption in developed societies, it seems reasonable to introduce fish oil in capsule supplement dosage forms and several food products enriched with fish oil that can be an additional source of the desirable long-chain omega-3 PUFA in the diet. For this purpose, reaching the recommended daily intake may require taking several capsules of fish oil per day.

Several studies have been performed to evaluate the potential health benefits brought by the consumption of food enriched with fish oil. Some studies suggest that different amounts of long-chain omega-3 - DHA and EPA, provided in a supplement form or added to food products, result in the same effect in changes in the blood lipid profile. The development of fish oil enriched food must be based on the scientific knowledge of the target function in the body and show that the effects are relevant for improved health or reduction of disease risk. The physiological effects of the intake of omega-3 fatty acids added to foods may differ depending on the quality of the fish oil used and the type of product.

Fish oil benefits range from decreasing risk of the so-called life-style diseases, particularly cardiovascular diseases, to combating depression, bipolar disorder and schizophrenia. Fish oil has also prophylaxis effects and treatment effects on inflammation, arthritis, anti-aging, age-related macular degeneration and mental health. Most of dietary lipids ingested from food consist of triacyglycerols. Prior to passive diffusion into the enterocytes, lipid digestion and emulsification are initiated by the action of different lipases resulting in the release of 2 free fatty acids and one monoglyceride-linked fatty acid. They are incorporated into mixed micelles to facilitate absorption into the bloodstream. The process of manufacturing the fish oil determines the quality which also depends on the type of fish used and the purity standards followed when refining the oil. Emulsified forms of fish oil have led to improved digestion and absorption of EPA and DHA in human healthy volunteers.

Flavored emulsified liquid preparations provide a simplified approach to fish oil delivery; emulsion as new approach seems to have advantages in the digestion and absorption of fatty acids which will increase the bioavailability. Using a novel approach of fish oil emulsification, preliminary results have indicated that both the rate and the extent of absorption of the fatty acids, particularly EPA and DHA, may be increased when digested. The present study was designed to establish that fish oil pre-emulsified using a novel approach will lead to increased absorption of EPA and DHA compared with the non-emulsified form of the fish oil.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged 18-60 years (inclusive Body mass index between 19 and 30 kg / m² (inclusive) at the pre-selection visit Individuals had to refrain from participating to other clinical studies involving experimental drugs for at least 30 days.

Female of childbearing potential must have an adequate contraception

Exclusion Criteria:

Person who consumed natural health products containing n-3 FAs in the last 6 months Allergy to fish or seafood Moderate-to-severe lipidemia (total cholesterol ≤ 240 mg/dl; LDL ≤ 160 mg/dl; Triglyceride ≤ 199 mg/dl) Tobacco or drug use Regular use of alcohol (females > 10 drinks, males > 14 drinks per week) Person who donated blood or had significant blood loss in the 56 days prior to study start Individuals with systolic blood pressure above 160 mmHg and diastolic blood pressure above 95 mmHg, or cardiac output at rest of less than 40 beats per minute or greater than 100 beats per minute.

People presenting any cardiovascular, pulmonary, haematological, neurological, psychiatric, endocrine or immunological problems as well as any gastrointestinal tract, liver, kidney disease or other conditions that could affect the absorption of lipids Hypothyroidism Positive human chorionic gonadotropin, a hormone secreted during pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-11-11 (Actual); Primary Completion 2011-03-31 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
The absorption of EPA and DHA in the plasma | 0-5 hours
  Define by the area under the curve between 0-5h
The bioavailability of EPA and DHA in the plasma | 0-24 hours
  Define by the area under the curve between 0-24h

SECONDARY OUTCOMES:
The maximum concentration of EPA and DHA in the plasma | 0-24 hours
  Define by the highest concentration achieved by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Plourde, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de Recherche sur le Vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No